CLINICAL TRIAL: NCT04845763
Title: Validation of the QoR-15 Score for Assessing Quality of Recovery From Emergency Surgery and Its Association With Long-term Quality of Life.
Brief Title: Validation of the QoR-15 Score for Emergency Surgery
Acronym: FQoR-15U
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: FQoR-15U
Record Dates: First submitted 2021-04-11; First posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Quality of Recovery; Perioperative Complication; Anesthesia; Patient Reported Outcome Measures; Surgery; Postoperative Complications; Emergency Surgery
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: Each patient complete the french version of the QoR-15 score (FQoR-15) at 3 times (before surgery, on Day 1, on Day 2).
  Interventions: Other: FQoR-15 questionnaire

INTERVENTIONS:
Other: FQoR-15 questionnaire — The FQoR-15 questionnaire (French version) consists of 15 questions concerning five domains (the patient's feelings, comfort, pain, dependence on the health care team and psychological well-being). Two to three minutes are required to complete all the questions. If the patient is not able to read the questionnaire himself, a third person can ask the patient the questions orally. In the case of ambulatory surgery, the patient is contacted by telephone to answer the questionnaire. Each item is scored from 0 to 10 and the total score is the sum of the score obtained for each item, i.e. a score from 0 to 150.

SUMMARY:
Recovery from surgery is a complex process, depending on the characteristics of the patient, the anesthesia used, and the time required for surgical management.

In the context of emergency surgery, the perioperative period is associated with an increase in morbidity and mortality, which may lead us to suspect an alteration in the quality of recovery.

Different scales to measure the quality of post-operative recovery have been developed. The QoR-40 and QoR-15 questionnaires assess recovery after elective surgery.These scoring tools accurately measure postoperative recovery by addressing key domains: pain, physical comfort, physical independence, psychological support and emotional state. Their use is recommended as an endpoint for assessing patient comfort in clinical trials, according to the Standardized Endpoints in Perioperative Medicine (StEP) initiative. In addition, monitoring of the QoR-15 is recommended by the American Society for Enhanced Recovery. A recent French translation of the QoR-15 score has been validated for use in scheduled surgery.

All of these scores, regardless of the language in which they are translated, have been developed and validated in patients who have undergone scheduled surgery. Until now, no validated scoring tool has been available to assess recovery after emergency surgery, whether traumatological or not.

DETAILED DESCRIPTION:
Recovery from surgery is a complex process, depending on the characteristics of the patient, the anesthesia used, and the time required for surgical management. This event is a source of stress, anxiety, pain, and even complications, both minor (nausea, vomiting) and major (such as surgical revision). The perioperative management and the psychological support allocated to each patient will have an impact on the hospitalization experience.

In the context of emergency surgery, the perioperative period is associated with an increase in morbidity and mortality, which may lead us to suspect an alteration in the quality of recovery.

Most clinical studies are interested in the reduction of perioperative morbidity and mortality (e.g. decrease in pain intensity measured by a visual analog scale, decrease in the frequency of nausea/vomiting, decrease in the time to remobilization, etc.) but still few of them evaluate in a global way the recovery, in particular in the emergency context.

Currently there is a desire to improve the physical and psychological recovery of our patients. In this context, scales to measure the quality of post-operative recovery have been developed. The QoR-40 and QoR-15 questionnaires assess recovery after elective surgery.These scoring tools accurately measure postoperative recovery by addressing key domains: pain, physical comfort, physical independence, psychological support and emotional state. Their use is recommended as an endpoint for assessing patient comfort in clinical trials, according to the Standardized Endpoints in Perioperative Medicine (StEP) initiative. In addition, monitoring of the QoR-15 is recommended by the American Society for Enhanced Recovery. A recent French translation of the QoR-15 score has been validated for use in scheduled surgery.

All of these scores, regardless of the language in which they are translated, have been developed and validated in patients who have undergone scheduled surgery. Until now, no validated scoring tool has been available to assess recovery after emergency surgery, whether traumatological or not.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old,
* French speaking,
* Admitted for any type of urgent surgery (time to surgery < 72 hours) traumaor not
* Able to answer the questionnaire at hospital admission, alone or with the help of a third party,
* And agreeing to participate in the study.

Exclusion Criteria:

* Patients with psychiatric or neurological pathologies that compromise cooperation with the protocol,
* Patients admitted for cardiac surgery or obstetrical surgery (caesarean section),
* Patients admitted for revision surgery,
* Patients already included in the study during a previous admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted for emergency surgery
Sampling Method: Non-Probability Sample
Enrollment: 375 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Validity of FQoR-15 questionnaire (24 hours) | At 24 hours after surgery
  Evaluate the validity of the French version of the QoR-15 to assess immediate postoperative recovery after emergency surgery (at 24 hours)
Validity of FQoR-15 questionnaire (48 hours) | At 48 hours after surgery
  Evaluate the validity of the French version of the QoR-15 to assess immediate postoperative recovery after emergency surgery (at 48 hours)

SECONDARY OUTCOMES:
Validity of FQoR-15 questionnaire for trauma surgery | At 24 and 48 hours after surgery
  Ensure the validity of the questionnaire in the sub-population of trauma emergency surgery at 24 and 48 hours
Validity of FQoR-15 questionnaire for non-traumatic surgery | At 24 and 48 hours after surgery
  Ensure the validity of the questionnaire in the sub-population of non-traumatic emergency surgery at 24 and 48 hours
Minimal important difference | At 24 and 48 hours after surgery
  Estimate minimal important difference from the FQoR-15 questionnaire in the emergency surgery population.
Quality of life (EQ5D-3L) | 3 months after surgery
  To study the association between the quality of postoperative recovery (both at 24 hours and at 48 hours of surgery) with quality of life at 3 months (measured by the EQ5D-3L visual analog scale)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leger M, Campfort M, Cayla C, Parot-Schinkel E, Lasocki S, Rineau E. Validation of an alternative French version of the Quality of Recovery-15 Score: the FQoR-15. Br J Anaesth. 2020 Oct;125(4):e345-e347. doi: 10.1016/j.bja.2020.05.052. Epub 2020 Jul 9. No abstract available. PMID 32654751
- [Derived] Le Bescond V, Petit-Phan J, Campfort M, Nicolleau C, Conte M, Bouhours G, Rony L, Lasocki S, Leger M. Validation of the postoperative Quality of Recovery-15 questionnaire after emergency surgery and association with quality of life at three months. Can J Anaesth. 2024 May;71(5):590-599. doi: 10.1007/s12630-024-02722-4. Epub 2024 Mar 19. PMID 38504036